CLINICAL TRIAL: NCT02246452
Title: Assessment of the Nutritional Status of Children and Adolescents With Malignancies Aged Between 0-18, Based on BMI Percentiles and Standard Deviation Scores, at Diagnosis, During Treatment, and During Two Years Follow-up
Brief Title: Assessment of the Nutritional Status of Children and Adolescents With Malignancies
Status: Completed | Type: Observational
Sponsor: University of Hohenheim (Other)
Collaborators: Olgahospital Stuttgart (Unknown)
Responsible Party: Sponsor
Other Study IDs: EM-13
Record Dates: First submitted 2014-09-17; First posted 2014-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Malnutrition
Keywords: Children and adolescents; Cancer; Malnutrition; BMI percentile; BMI-SDS
MeSH Terms: conditions — Malnutrition; Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective of this study was the assessment of the nutritional status of children and adolescents aged between 0-18 with malignancies based on BMI percentiles and standard deviation scores, at diagnosis, during treatment and during a period of two years after the end of therapy.

DETAILED DESCRIPTION:
Children and adolescents suffering from malignancies often show malnutrition. Malnutrition, defined as a deficiency or an excess of energy, is associated with an increased risk of comorbidities, reduced survival rates, higher relapse rates, and worse treatment response.

The present retrospective study assessed the nutritional status of children and adolescents, suffering from nine different kinds of cancer, based on BMI percentiles and standard deviation scores. Anthropometric data were recorded from clinical charts and an assessment of the nutritional status was made at the beginning of treatment, during the course of therapy and during a follow-up period of two years. The influence of treatment-related characteristics, the duration of therapy, and the occurrence of a relapse or progress during therapy on the nutritional status were examined.

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents treated at the Olgahospital Stuttgart for one of the nine different cancer types
* treated according to a study protocol of the Society of Pediatric Oncology and Hematology (GPOH), with modifications only allowed within the therapeutic protocol
* time period between diagnosis and start of treatment less than 28 days
* age younger than 18

Exclusion Criteria:

* severe underlying disease, which exerts a strong influence on weight and/or height
* patients whose clinical record does not state any weight and/or height
* diseases which are not considered as malignant because of the state or biology

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents, treated for one of the following diseases: lymphoma, germ cell tumor, nephroblastoma, soft tissue sarcoma, neuroblastoma, Ewing sarcoma, brain tumor, or acute lymphoblastic leukemia (ALL)/acute myeloid leukemia (AML)
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Nutritional status at diagnosis | Within the month of diagnosis
  To assess the nutritional status height and weight were recorded from patient charts to calculate the BMI percentile (Body Mass Index percentile) and the BMI-SDS (Body Mass Index-Standard Deviation Score)
Change in nutritional status during treatment | Every month during the treatment period (average treatment period 11 months)
  To assess the nutritional status height and weight were recorded from patient charts to calculate the BMI percentile and the BMI-SDS
Change in nutritional status during follow-up | Once in a period of three months during two years follow-up
  To assess the nutritional status height and weight were recorded from patient chart to calculate the BMI percentile and the BMI-SDS

SECONDARY OUTCOMES:
Clinical picture | Within the month of diagnosis
  Kind of cancer (lymphoma, germ cell tumor, nephroblastoma, soft tissue sarcoma, neuroblastoma, Ewing sarcoma, brain tumor, acute lymphoblastic leukemia (ALL)/acute myeloid leukemia (AML)), recorded from patient chart
Age (years) | Within the month of diagnosis
  Age in years, recorded from patient chart
Treatment period (months) | Patients were followed for the duration of their treatment period. Average treatment period 11 months
  Time from start until the end of treatment, recorded from patient chart
Incidence of nutritional interventions | Patients were followed for the incidence of a nutritional intervention within the treatment period (average treatment period 11 months)
  Application of parenteral nutrition or gastric tube (yes/no), recorded from patient chart
Infection | Patients were followed for the occurence of an infection within the treatment period (average treatment period 11 months)
  Occurence of an infection (yes/no), recorded from patient chart
Fever | Patients were followed for the occurence of fever within the treatment period (average treatment period 11 months)
  Occurence of fever (yes/no), recorded from patient chart
Administration of antibiotics | Patients were followed for the occurence of an administration of antibiotics within the treatment period (average treatment period 11 months)
  Administration of antibiotics (yes/no), recorded from patient chart
Diarrhea | Patients were followed for the occurence of diarrhea within the treatment period (average treatment period 11 months)
  Occurence of diarrhea (yes/no), recorded from patient chart
Mucositis | Patients were followed for the occurence of mucositis within the treatment period (average treatment period 11 months)
  Occurence of mucositis (yes/no),recorded from patient chart
Nausea | Patients were followed for the occurence of nausea within the treatment period (average treatment period 11 months)
  Occurence of nausea (yes/no), recorded from patient chart
Constipation | Patients were followed for the occurence of constipation within the treatment period (average treatment period 11 months)
  Occurence of constipation (yes/no), recorded from patient chart
Relapse/Progress | Patients were followed for the occurence of a relapse/progress within the treatment period (average treatment period 11 months) and follow-up (two years)
  Occurence of a relapse/progress (yes/no), recorded from patient chart
Kind of treatment | Patients were followed for the kind of treatment they received wihin the treatment period (average treatment period 11 months)
  Kind of treatment (chemotherapy, operation, Radiation), recorded from Patient chart